CLINICAL TRIAL: NCT04053998
Title: Benchmarking Outcomes in Pancreatoduodenectomy With Portal Vein Resection - WhippleBenchmarks.Org
Brief Title: Benchmarking Outcomes in Pancreatic Surgery - WhippleBenchmarks.Org
Status: Completed | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Cancer Institute Hospital, Japan (Other); Hospital Curry Cabral, CHLC, Lisbon, Portugal (Unknown); St. Joseph's Hospital of Atlanta (Other); Erasmus Medical Center (Other); Hospital Italiano de Buenos Aires (Other); Juntendo University (Other); Parc de Salut Mar (Other); Queen Elizabeth Hospital NHS Foundation Trust (Other); Rennes University Hospital, Rennes, France (Unknown); San Raffaele University Hospital, Italy (Other); St Vincent's University Hospital, Ireland (Other); Thomas Jefferson University (Other); University of Dublin, Trinity College (Other); University of Lyon (Other); Mainz University (Other); University of Pisa (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); University Hospital Southampton NHS Foundation Trust (Other); University Hospital, Zürich (Other); Amsterdam UMC, location VUmc (Other); University of Colorado, Denver (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Dimitri Raptis, Senior Clinical Fellow in HPB and Transplant Surgery, Royal Free Hospital NHS Foundation Trust
Other Study IDs: WB-08-2019
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Pancreatic Neoplasms; Pancreaticoduodenectomy
Keywords: Pancreaticoduodenectomy; Portal vein resection; Benchmarks; Outcomes
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy with portal vein resection — Pancreatic surgery with vein resection to achieve disease clearance.

SUMMARY:
The WhippleBenchmark 2 Collaborative study aims at defining benchmark criteria for best achievable outcomes after pancreaticoduodenectomy with portal vein resection.

DETAILED DESCRIPTION:
Pancreatoduodenectomy (PD) with portal vein resection (PVR) is performed for the achievement of complete resection (R0) in patients with locally advanced pancreatic head lesions. Despite most commonly performed in high-volume pancreatic surgery centers by experienced surgeons, best achievable outcomes, such as morbidity and mortality, following such complex procedure remain unknown.

The aim is to conduct a retrospective multicenter cohort study to define benchmark values for best achievable outcomes following duodenopancreatectomy (DP) with portal vein resection (PVR).

Data collection and study design are based on to the well established standardized reporting for benchmarking (Sánchez-Velázquez et. al. Ann Surg, February 2019 ).

This multicenter cohort study will include all consecutive pancreaticoduodenectomies with portal vein resections from at least 20 high volume centers performing over 50 pancreatic operations per year or 150 cases within 3 years from at least 3 continents over a period of 10 years (2009-2019). Every center included in the study must have a prospective database from which data can be collected as well as previous publications critically reporting on their outcome.

ELIGIBILITY:
Center Eligibility Criteria

* High volume centers from ≥3 continents
* Minimum 50 cases of pancreatic surgery per year or 150 cases within 3 years
* Published in the area of pancreas surgery
* Prospective database available

Patient Eligibility Criteria

Inclusion Criteria:

* Adults ≥ 18 years
* Resectable malignant or benign diseases (i.e. all indications)
* Open pancreaticoduodenectomy (all techniques allowed) with concurrent portal vein resection

Exclusion Criteria:

* Patients < 18 years
* Pancreatic resections other than pancreaticoduodenectomy and portal vein resection
* Pancreaticoduodenectomy with arterial reconstruction
* Laparoscopic or robotic pancreaticoduodenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic malignancy that underwent open pancreaticoduodenectomy with portal vein resection.
Sampling Method: Non-Probability Sample
Enrollment: 1462 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 12 months
  Death due to any cause postoperatively
Morbidity rate | 12 months
  Classified according to the Clavien-Dindo Classification of postoperative complications.
Morbidity assessed according to the Comprehensive Complications Index® (CCI®) | 12 months
  The Comprehensive Complications Index® (CCI®) reports the cumulative postoperative morbidity, a novel metric which measures the overall morbidity on a scale from 0 (no complications) to 100 (death).

SECONDARY OUTCOMES:
Pancreatic fistula rates | 12 months
  reported according to both the International Study Group of Pancreatic Fistula (ISGPF) and Clavien-Dindo classification.
Hospital readmission rate | 12 months
  Any hospital readmission to the primary or other peripheral hospitals
Disease free survival rate | Up to 10 years postoperatively
  Disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe K Fusai, MD, Principal Investigator — Royal Free Hospital, London, UK; Dimitri A Raptis, MD, MSc, PhD, Principal Investigator — Royal Free Hospital, London, UK; Patricia Sánchez Velázquez, MD, PhD, Principal Investigator — Parc de Salut Mar, Barcelona, Spain; Nikolaos Machairas, MD, Principal Investigator — Royal Free Hospital, London, UK
Locations (2):
- Parc de Salut Mar, Barcelona, Spain
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study Investigators will act as the custodians of the data. The data however belong to all collaborators. The study investigators will decide after the publication of the main report about requests from the collaborators regarding secondary analyses and will consider all such requests based on quality and the validity of the proposed project.
Supporting Information: Study Protocol
Time Frame: The data will remain available to share with the collaborators as described above up to 5 years after the study completion.
Access Criteria: Quality and validity of the proposed project.
URL: https://whipplebenchmarks.org

REFERENCES:
- [Background] Sanchez-Velazquez P, Muller X, Malleo G, Park JS, Hwang HK, Napoli N, Javed AA, Inoue Y, Beghdadi N, Kalisvaart M, Vigia E, Walsh CD, Lovasik B, Busquets J, Scandavini C, Robin F, Yoshitomi H, Mackay TM, Busch OR, Hartog H, Heinrich S, Gleisner A, Perinel J, Passeri M, Lluis N, Raptis DA, Tschuor C, Oberkofler CE, DeOliveira ML, Petrowsky H, Martinie J, Asbun H, Adham M, Schulick R, Lang H, Koerkamp BG, Besselink MG, Han HS, Miyazaki M, Ferrone CR, Fernandez-Del Castillo C, Lillemoe KD, Sulpice L, Boudjema K, Del Chiaro M, Fabregat J, Kooby DA, Allen P, Lavu H, Yeo CJ, Barroso E, Roberts K, Muiesan P, Sauvanet A, Saiura A, Wolfgang CL, Cameron JL, Boggi U, Yoon DS, Bassi C, Puhan MA, Clavien PA. Benchmarks in Pancreatic Surgery: A Novel Tool for Unbiased Outcome Comparisons. Ann Surg. 2019 Aug;270(2):211-218. doi: 10.1097/SLA.0000000000003223. PMID 30829701
- [Background] Raptis DA, Mettler T, Fischer MA, Patak M, Lesurtel M, Eshmuminov D, de Rougemont O, Graf R, Clavien PA, Breitenstein S. Managing multicentre clinical trials with open source. Inform Health Soc Care. 2014 Mar;39(2):67-80. doi: 10.3109/17538157.2013.812647. PMID 24517456
- [Derived] Raptis DA, Sanchez-Velazquez P, Machairas N, Sauvanet A, Rueda de Leon A, Oba A, Groot Koerkamp B, Lovasik B, Chan C, Yeo CJ, Bassi C, Ferrone CR, Kooby D, Moskal D, Tamburrino D, Yoon DS, Barroso E, de Santibanes E, Kauffmann EF, Vigia E, Robin F, Casciani F, Burdio F, Belfiori G, Malleo G, Lavu H, Hartog H, Hwang HK, Han HS, Poves I, Rosado ID, Park JS, Lillemoe KD, Roberts KJ, Sulpice L, Besselink MG, Abuawwad M, Del Chiaro M, de Santibanes M, Falconi M, D'Silva M, Silva M, Abu Hilal M, Qadan M, Sell NM, Beghdadi N, Napoli N, Busch ORC, Mazza O, Muiesan P, Muller PC, Ravikumar R, Schulick R, Powell-Brett S, Abbas SH, Mackay TM, Stoop TF, Gallagher TK, Boggi U, van Eijck C, Clavien PA, Conlon KCP, Fusai GK. Defining Benchmark Outcomes for Pancreatoduodenectomy With Portomesenteric Venous Resection. Ann Surg. 2020 Nov;272(5):731-737. doi: 10.1097/SLA.0000000000004267. PMID 32889866
- See also: rBiostatistics.com - Cloud Graphical User Interface for R Statistics and eLearning Platform — https://rBiostatistics.com
- See also: The Comprehensive Complications Index® (CCI®) — https://www.assessurgery.com